CLINICAL TRIAL: NCT03742024
Title: Observational Study of Pediatric Migraine: The Pediatric Migraine Registry
Brief Title: Study of Pediatric Migraine: The Pediatric Migraine Registry
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00100205
Record Dates: First submitted 2018-11-12; First posted 2018-11-15 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Months
Biospecimen Retention: Samples With DNA — Whole blood, buccal swab, urine, stool.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children and adolescents: Children and adolescents between the ages of 4 and 17 years old (inclusive)

SUMMARY:
This is a multi-center registry that will prospectively collect regulatory compliant data from children and adolescents with migraine. This study will enroll approximately 200 participants from approximately 20 sites and will examine migraine symptoms, therapeutics used, and biomarkers associated with migraine.

ELIGIBILITY:
Inclusion Criteria:

* 4 to 17 years of age inclusive at the time of enrollment visit
* Meets International Classification of Headache Disorders, 3rd edition criteria for migraine with or without aura
* Guardian provides informed consent/HIPAA
* Participant provides assent if developmentally appropriate and required by the institutional review board

Exclusion Criteria:

* Any condition which would make the participant, in the opinion of the investigator, unsuitable for the study

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Participants aged 4-17 years old (inclusive) diagnosed with migraine with or without aura will be eligible for participation in this study.
Sampling Method: Non-Probability Sample
Enrollment: 201 (Actual)
Dates: Start 2018-12-05 (Actual); Primary Completion 2021-02-08 (Actual); Study Completion 2021-02-08 (Actual)

PRIMARY OUTCOMES:
Migraine frequency | Approximately 12 months
  Number of days per month participant experiences migraine

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Hornik, MD, Principal Investigator — Duke University; Amy Gelfand, MD, Principal Investigator — University of California at San Francisco
Locations (19):
- United States (19):
  - University of California at San Francisco, San Francisco, California
  - Colorado Springs Neurological Associates, Colorado Springs, Colorado
  - Nemours Alfred I duPont Hospital For Children Neurology, Wilmington, Delaware
  - Nicklaus Children's Hospital, Miami, Florida
  - University of Louisville Health Sciences center, Louisville, Kentucky
  - University of Maryland, Baltimore, Maryland
  - Michigan Headache & Neurological Institute, Ann Arbor, Michigan
  - Children's Mercy Hospital, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Akron Children's Hospital, Akron, Ohio
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - The Cleveland Clinic Children's Hospital, Cleveland, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Rhode Island Hospital, The Miriam Hospital, Providence, Rhode Island
  - University of South Carolina at Columbia, Columbia, South Carolina
  - University of Vermont School of Medicine, Burlington, Vermont
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No